CLINICAL TRIAL: NCT02428218
Title: A Randomized, Placebo-Controlled, Parallel-Group Study in Pediatric Subjects Ages 10 Through 17 Years to Evaluate the Efficacy and Safety of BG00012 for the Treatment of Relapsing-Remitting Forms of Multiple Sclerosis
Brief Title: Placebo-Controlled Study of the Efficacy and Safety of BG00012 in Pediatric Subjects With Relapsing-Remitting Multiple Sclerosis (RRMS)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Feasibility
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109MS309; 2014-005624-98 (EudraCT Number)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Relapsing Forms of Multiple Sclerosis
Keywords: Randomized; Ages 10-17; Pediatrics; Placebo controlled; Relapse-Remitting; Multiple Sclerosis; Safety; Efficacy; BG00012
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BG00012 (Experimental): Participants will receive 120 mg capsule(s) BG00012 taken orally.
  Interventions: Drug: dimethyl fumarate
- Placebo (Experimental): Participants will receive matching placebo capsule(s) taken orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dimethyl fumarate — enteric-coated microtablets
  Other Names: BG00012; DMF
  Arms: BG00012
Drug: Placebo — enteric-coated microtablets
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of oral BG00012 as compared with placebo in pediatric subjects with relapsing-remitting multiple sclerosis (RRMS). The secondary objectives of this study are to evaluate the safety and tolerability of BG00012 and to compare the effect of BG00012 with placebo on additional clinical and radiological measures of disease activity.

ELIGIBILITY:
Key Inclusion Criteria:

* Informed consent and assent as appropriate
* Must have a body weight of ≥30 kg
* Must have a diagnosis of RRMS as defined by the revised consensus definition for pediatric multiple sclerosis (MS)
* Must be ambulatory with a converted Krutzke Baseline Expanded Disability Status Scale (EDSS) score between 0 and 5.0, inclusive

Key Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS.
* History of disorders mimicking MS, such as other demyelinating disorders (e.g., acute disseminated encephalomyelitis), systemic autoimmune disorders (e.g., Sjögren disease and lupus erythematosus), metabolic disorders (e.g., dystrophies), and infectious disorders.
* History of severe allergic or anaphylactic reactions, or known drug hypersensitivity to dimethyl fumarate (DMF) or fumaric acid esters.
* Prior treatment with any of the following medications within 12 months prior to randomization: mitoxantrone, cyclophosphamide, rituximab.
* Prior treatment with any of the following medications or procedures within 6 months prior to randomization: fingolimod, teriflunomide, natalizumab, cyclosporine, azathioprine, methotrexate, mycophenolate mofetil, laquinimod, intravenous (IV) immunoglobulin, plasmapheresis or cytapheresis.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time to first multiple sclerosis (MS) relapse | Up to week 104
  Relapses are defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Examining Neurologist.

SECONDARY OUTCOMES:
Number of participants that experience adverse events (AEs) and serious adverse events (SAEs) | Up to week 104
Number of new or newly enlarging T2 Hyperintense Lesions on Brain magnetic resonance imaging (MRI) scans | Weeks 24, 48, 72 and 96
Number of gadolinium-enhancing Lesions | Baseline, and weeks 24, 48, 72 and 96
Annualized MS relapse rate | weeks 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen